CLINICAL TRIAL: NCT05150210
Title: A Prospective, Multi-Center Investigation of the da Vinci SP Surgical System in Pulmonary and Lobectomy for Benign and Malignant Disease
Brief Title: SP Thoracic IDE Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SP Thoracic IDE
Record Dates: First submitted 2021-11-24; First posted 2021-12-09 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-09

CONDITIONS: Primary Lung Cancer; Benign Lung Disease; Thymoma; Myasthenia Gravis
MeSH Terms: conditions — Thymoma; Myasthenia Gravis | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SP Surgical System- Lobectomy procedures (Experimental): Pulmonary lobectomy performed by da Vinci SP Surgical System.
  Interventions: Device: Robotic-Assisted Surgery
- SP Surgical System - Thymectomy (Experimental): Thymectomy procedures performed by the da Vinci SP Surgical System
  Interventions: Device: Robotic-Assisted Surgery

INTERVENTIONS:
Device: Robotic-Assisted Surgery — da Vinci SP Surgical System, instruments, and accessories in pulmonary lobectomy and thymectomy for benign and malignant disease.

SUMMARY:
To confirm the safety and performance of the da Vinci SP Surgical System, Instruments and Accessories in pulmonary lobectomy, and in thymectomy procedures.

DETAILED DESCRIPTION:
Primary performance:

The primary endpoint will be assessed as the ability to complete the planned da Vinci SP-assisted thoracic procedure without conversion to an alternate approach. Conversion to an alternate approach comprises undocking of the da Vinci SP to complete the planned procedures using other methods, such as open, VATS, or multiport robotic (da Vinci SI or X/Xi)

Primary Safety:

The primary safety endpoint will be assessed as the incidence of all intra-operative and post-operative adverse events that occur through the 30-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* BMI ≤ 35
* ASA ≤ 3
* Willing and able to provide a written informed consent
* Willing and able to comply with the study protocol requirements including follow-up examinations at 14 days and 30 days post-operatively, and post-market long term follow-up on an annual basis through 5 years

Lobectomy Inclusion Criteria:

- Clinical stage I or II primary lung cancer or other suspected lung malignancy; or benign lung disease requiring resection; primary tumor ≤ 5cm diameter

Thymectomy Inclusion Criteria:

- Masaoka clinical stage I or II thymoma; or thymectomy for myasthenia gravis; thymic mass ≤ 5 cm diameter

Exclusion Criteria:

* Clinical or radiological evidence of mediastinal or systemic metastatic disease
* Life expectancy < 6 months
* Subject with a known bleeding or clotting disorder
* Subjects actively receiving therapeutic-dose anticoagulation or anti-platelet medications at the time of operation
* Uncontrolled systemic illness 6 months prior to planned surgical procedure including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Previous chemotherapy, immunotherapy and/or radiation therapy for treatment of the cancer to be resected
* Subject has a contraindication for general anesthesia or surgery
* Subjects under active immunomodulatory or immunosuppressive regimen (e.g. transplant patient, high-dose steroid requirement) within 30 days prior to the planned surgical procedure. For myasthenia patients, if steroids are weaned down to prednisone ≤ 5 mg/day prior to day of surgery, the patient may be enrolled
* Previous sternotomy
* Subject belongs to vulnerable population
* Subject is pregnant or suspected to be pregnant or breastfeeding

Lobectomy Exclusion Criteria:

* Tumor involving carina or any airway requiring sleeve resection, bronchoplasty
* Tumor requiring resection of local structures (e.g. chest wall) or extended resection such as bilobectomy
* History of pulmonary hypertension
* Previous ipsilateral thoracic surgery or radiotherapy

Thymectomy Exclusion Criteria:

* Uncontrolled myasthenia gravis symptoms at the time of scheduled surgery
* Tumor requiring resection of local structures (except pericardium)
* Confirmed thymic carcinoma

Intraoperative Exclusion Criteria:

- Anatomy determined intra-operatively to be unsuitable for minimally invasive surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2028-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Rice, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SP Surgical System -Thymectomy: Thymectomy procedures performed by da Vinci SP Surgical System.
- SP Surgical System - Lobectomy: Lobectomy procedures performed by the SP Surgical System
Period: Overall Study
Arm/Group | SP Surgical System -Thymectomy | SP Surgical System - Lobectomy
Started | 13 | 19
Completed | 13 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SP Surgical System - Thymectomy: Pulmonary thymectomy procedures performed by da Vinci SP Surgical System.
- SP Surgical System - Lobectomy: Pulmonary lobectomy procedures performed by da Vinci SP Surgical System.
- Total: Total of all reporting groups
Arm/Group | SP Surgical System - Thymectomy | SP Surgical System - Lobectomy | Total
Number analyzed (Participants) | 13 | 19 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Thymectomy and Lobectomy groups were analyzed separately, including analysis for Age.
  years
    Thymectomy: number analyzed (Participants) | 13 | 0 | 13
    Thymectomy | 54.5 (15.86) |  | 54.5 (15.86)
    Lobectomy: number analyzed (Participants) | 0 | 19 | 19
    Lobectomy |  | 66.4 (8.06) | 66.4 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 2 | 13 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 12 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Conversion
Description: Performance defined as the ability to complete the planned da Vinci SP-assisted pulmonary lobectomy and thymectomy procedures without conversion to an alternate approach
Time Frame: Intra-operative period
Population: 0 Conversions occured
Measure: Count of Participants; unit: Participants
Groups:
- SP Surgical System- Thymectomy Arm: Thymectomy procedures performed by da Vinci SP Surgical System.
- SP Surgical System - Lobectomy Arm: Lobectomy procedures performed by the da Vinci SP Surgical System.
Arm/Group | SP Surgical System- Thymectomy Arm | SP Surgical System - Lobectomy Arm
Number analyzed (Participants) | 13 | 19
Participants | 0 | 0

2. Primary Outcome: Major Adverse Event Rate
Description: Safety defined as the incidence of major intra-operative and post-operative adverse events that occur through the 30-day follow-up period.
Time Frame: Intra-operative through the 30 days follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | SP Surgical System- Thymectomy Arm | SP Surgical System - Lobectomy Arm
Number analyzed (Participants) | 13 | 19
Participants | 0 | 3

ADVERSE EVENTS:
Time Frame: Through the 30 day follow up period.
Description: Major adverse events: Clavien-Dindo Grade III or higher
Groups:
- SP Surgical System- Thymectomy: Thymectomy procedures performed by da Vinci SP Surgical System.
- SP Surgical System- Pulmonary Lobectomy: Pulmonary lobectomy procedures performed by da Vinci SP Surgical System.
Arm/Group | SP Surgical System- Thymectomy | SP Surgical System- Pulmonary Lobectomy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/13 | 4/19
Other Adverse Events (participants affected / at risk) | 5/32 | 5/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SP Surgical System- Thymectomy (N=13) | SP Surgical System- Pulmonary Lobectomy (N=19)
Air Leakage (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SP Surgical System- Thymectomy (N=32) | SP Surgical System- Pulmonary Lobectomy (N=19)
Intraoperative Adverse Event (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Non-serious AE (General disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT05150210/Prot_SAP_001.pdf